CLINICAL TRIAL: NCT05650840
Title: Enamel Abrasion and Stain Removal Efficacy of Charcoal -Based and Calcium Carbonate /Perlite Whitening Toothpastes: A Randomized Clinical Trial and In-vitro Trial
Brief Title: Enamel Abrasion and Stain Removal Efficacy of Two Whitening Toothpastes: An In-vitro and In-vivo Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Osama Metwally, Master student, conservative department, faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU-2022
Record Dates: First submitted 2022-11-24; First posted 2022-12-14 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Tooth Abrasion
Keywords: Charcoal based toothpaste; External tooth stains; Teeth abrasion
MeSH Terms: conditions — Tooth Abrasion | interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Charcoal -based whitening toothpaste (Experimental): signal charcoal white& Detox toothpaste Unilever Mashreq - Egypt
  Interventions: Procedure: Charcoal based whitening toothpaste (signal charcoal white& Detox toothpaste Unilever Mashreq - Egypt
- Calcium carbonate /perlite containing whitening toothpaste (Active Comparator): signal whitening moonlight toothpaste Unilever Mashreq - Egypt
  Interventions: Procedure: Calcium carbonate /perlite containing whitening toothpaste (signal whitening moonlight toothpaste Unilever Mashreq - Egypt).

INTERVENTIONS:
Procedure: Charcoal based whitening toothpaste (signal charcoal white& Detox toothpaste Unilever Mashreq - Egypt — The labial surface of anterior teeth will be brushed by the circular brushing technique twice daily (morning and after 6 hours) for at least 1 minute using charcoal containing toothpaste. Soft bristles toothbrushes will provided to all patients (Oral-B). After 1 month, re-evaluation of the stains will be performed and the data will be recorded.
  Intervention drug : whitening toothpaste charcoal based whitening toothpaste compared to calcium carbonate and perlite whitening toothpaste
  FOR IN VITRO:
  Human premolars will be obtained from volunteers due to orthodontic reasons. Teeth will be divided into two equal groups (n:18) according to the toothpaste used. Teeth will be brushed with an electric tooth brush (Oral-B PRO 500) that will be held in a holder to standardize the position to the tooth surface for 3 minutes equivalent to 2 times a day for one month. Teeth will be prepared for AFM examination
  Arms: Charcoal -based whitening toothpaste
Procedure: Calcium carbonate /perlite containing whitening toothpaste (signal whitening moonlight toothpaste Unilever Mashreq - Egypt). — The labial surface of anterior teeth will be brushed by the circular brushing technique twice daily (morning and after 6hours) for at least 1 minute using calcium carbonate /perlite containing toothpaste. Soft bristles toothbrushes will provided to all patients (Oral-B). After 1 month, re-evaluation of the stains will be performed and the data will be recorded. The main operator will perform the tooth brushing procedures for all the patients himself twice daily.
  FOR IN VITRO:
  Human premolars will be obtained from volunteers due to orthodontic reasons. Teeth will be divided into two equal groups (n:18) according to the toothpaste used. Teeth will be brushed with an electric tooth brush(Oral-B PRO 500) that will be held in a holder to standardize the position to the tooth surface for 3 minutes equivalent to 2 times a day for one month. Teeth will be prepared for AFM examination Device used is atomic force microscopy to determine enamel abrasion after brushing
  Arms: Calcium carbonate /perlite containing whitening toothpaste

SUMMARY:
The aim of the study is to clinically evaluate the efficacy of external stain removal of an activated charcoal based tooth paste versus calcium carbonate /perlite tooth paste. Additionally, to investigate enamel surface abrasion for both toothpastes in vitro.

DETAILED DESCRIPTION:
Statement of the problem:

Access to in-office treatments is restricted to a lot of population. Therefore, there has been an interest in developing methods so that patients can remove stains and apply tooth whitening at home. Accordingly, toothpastes, due to their ease of use and low cost, have been used as vehicles for whitening agents as an alternative to home/office whitening.

Hydrogen peroxide is the most commonly used agent for whitening teeth, which is used in various concentrations according to various techniques at home and office. Bleaching of teeth in office is done at a high concentration of Hydrogen peroxide for a specified period of time. In addition to conventional whitening treatments, over-the-counter products, including gels, toothpastes, bleaching strips, mouthwashes, and pens with different Hydrogen peroxide levels, have been developed. In-office teeth whitening is one of the more costly forms of teeth whitening and the concentration of the bleaching element is higher, it is better monitored by a professional.

Whitening toothpaste is probably the one of the most affordable options for someone looking to whiten their teeth at home, which contain abrasive and chemical agents and have the ability to remove external stains from the tooth. The abrasiveness of toothpastes depends on the hardness, size, and shape of abrasive particles. Furthermore, factors such as the brushing technique, brushing pressure, toothbrush hardness, and the number of brush strokes affect tooth abrasion. Abrasive agents include silica, phosphates, carbonates, and bicarbonates. Chemical agents present in whitening toothpastes are sodium citrate, phosphate salt. which react with chromogenic molecules of superficial dental stains and eliminate them from the tooth surface.

Whitening toothpastes include different active ingredients in their composition. It normally contain a higher amount of abrasives and detergents than do conventional toothpastes. In this sense, it is important to point out that toothpastes with higher amounts of abrasives may produce increased surface roughness in dental tissues, or restorations, or even tooth sensitivity, especially if they are used routinely.

Rationale:

Today, active charcoal is added to toothpastes which are marketed as charcoal toothpastes. The first report on the use of charcoal in oral and dental hygiene has been attributed to Hippocrates in ancient Greece. Charcoal is used as powder, soot, coal, and ash in different countries. Charcoal-based products are used in medical treatments, such as its use as an antidote for acute poisoning, drug overdose, skin infections. Charcoal is used legally for the coloring of food in China, Japan, and Korea to improve health.

Activated charcoal is produced as a natural method of the partial oxidation of various materials. High-porosity activated charcoal has the ability to exchange ion in the mouth through nanopores and can attach to tooth enamel and remove tooth-coloring agents (because of its capacity of adsorbing pigments, chromophores, and stains from the tooth surface). The application of this product has been suggested to eliminate some dental coloring agents. Charcoal can help tooth whitening through tooth abrasion.

ELIGIBILITY:
IN VIVO:

Patients inclusion:

* Adult male and female patients ≥18 years.
* Good oral and general health and oral hygiene have at least eight natural anterior teeth (incisors and canines) assessable for extrinsic stain and be available for all study appointments.

Patients exclusion:

* Uncooperative behavior.
* Patients allergic to tooth paste material.
* Patient with history of medical disease, drug therapies or any other serious relevant problem.
* Pregnant or breastfeeding women.
* Patients with fixed orthodontic appliances
* Patients who had professional tooth whitening, within the last six months.
* Patients who had significant amounts of calculus on facial surfaces of the incisors/canines.
* Patients who had undergone professional periodontal treatment within the previous six months or used mouth rinses for the treatment/ control of a periodontal condition.
* Patients who had advanced periodontal disease on anterior teeth.
* Xerostomic patients.
* Patients who used medications which could affect saliva flow or cause staining.
* Patients who had undergone dental prophylaxis within 8 weeks of screening.
* Patients who used minocycline or doxycycline within 30 days of screening or between screening and baseline.

Tooth inclusion:

▪ Vital anterior maxillary and mandibular teeth free of caries or restorations, no cervical lesions and no periodontal disease.

Tooth exclusion:

* Intrinsically Discolored teeth caused by tetracycline, fluorosis, hypocalcification hyperplasia, endodontic treatment (or requiring endodontic treatment).
* Restorations in anterior teeth, parafunctional habits or tooth sensitivity.
* Non- vital teeth.

IN-VITRO:

Teeth inclusion criteria:

* Intact, free of caries or restorations.
* No cervical lesions

Teeth exclusion criteria:

* Intrinsically Discolored teeth caused by tetracycline, fluorosis, hyperplasia, endodontic treatment .
* Restorations in teeth.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Stain scores as per Macpherson modification of the Lobene stain index | Baseline
  Stain scores will be recorded as per the Macpherson modified Lobene Stain Index area x intensity (AXI). Each tooth will be divided into four areas for assessment: gingival, mesial, distal and body. The stain index will measure area and intensity of extrinsic tooth stain on the facial surfaces of the anterior teeth.
  The criteria and codes for intensity were:
  0: no stain present, natural tooth colouration
  1. faint stain
  2. clearly visible stain, orange to brown (moderate stain)
  3. dark stain, deep brown to black (heavy stain) The area (extent) of the stain was recorded only if an intensity score was of 2 or 3
  The area criteria and codes for approximal and gingival sites were:
  1. thin line, can be continuous (< 1/3)
  2. thick line or band (>1/3, <2/3)
  3. covering total area (> 2/3)
Stain scores as per Macpherson modification of the Lobene stain index | after four weeks
  Stain scores will be recorded as per the Macpherson modified Lobene Stain Index area x intensity (AXI). Each tooth will be divided into four areas for assessment: gingival, mesial, distal and body. The stain index will measure area and intensity of extrinsic tooth stain on the facial surfaces of the anterior teeth.
  The criteria and codes for intensity were:
  0: no stain present, natural tooth colouration
  1. faint stain
  2. clearly visible stain, orange to brown (moderate stain)
  3. dark stain, deep brown to black (heavy stain) The area (extent) of the stain was recorded only if an intensity score was of 2 or 3
  The area criteria and codes for approximal and gingival sites were:
  1. thin line, can be continuous (< 1/3)
  2. thick line or band (>1/3, <2/3)
  3. covering total area (> 2/3)

OTHER OUTCOMES:
enamel abrasion using atomic force microscopy before and after brushing (Anton Paar - Tosca™ 200 - atomic force microscope, USA.) | 3 minutes equivalent to 2 times a day for one month
  evaluation the surface roughness of enamel before and after brushing using atomic force microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Iman I ElSayad, Study Director — Cairo University; Mohamed R El-Bialy, Post Phd, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No